CLINICAL TRIAL: NCT06556628
Title: Disco Thermometer Engineering Study Protocol
Brief Title: Tympanic Thermometer Study
Status: Active, not recruiting | Type: Observational
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 60117201
Record Dates: First submitted 2024-08-12; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Body Temperature Changes; Fever
MeSH Terms: conditions — Body Temperature Changes; Fever

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Fever: Elevated oral temperature of 37.5C or higher or elevated axillary temperature of 37.2C or higher.
  Interventions: Device: Increased Body Temperatures
- Healthy: Oral temperature between 36-37.4C Axillary temperature between 36-37.1C
- Cold: Oral or axillary temperatures below 36C

INTERVENTIONS:
Device: Increased Body Temperatures — Collecting data on patients whose body temperatures increase due to fighting an illness.
  Groups: Fever

SUMMARY:
The goal of this study is to collect febrile, healthy, and in some instances cold temperature data from human subjects ranging from newborns to geriatrics. This data will be used to develop a new thermometer.

ELIGIBILITY:
Inclusion Criteria:

* Age: normal weight (≥2.5kg), full-term (37 weeks gestation) newborn to geriatric adult.
* Participant, legal guardian, or healthcare proxy is able to give consent to participate.
* Participant, legal guardian, or healthcare proxy speaks fluent English.

Exclusion Criteria:

* The subject does not meet the inclusion criteria.
* The subject has anatomical abnormalities that would affect temperature.
* The subject has blood or drainage in the external ear canal.
* The subject has had something in their ear for a prolonged period, such as a hearing aid or headphones. The subject may be included if the hearing aid or headphones are removed at least 30 minutes prior to taking ear temperature.
* The subject has been lying on ear within 30 minutes of data collection. The subject may be included if they wait 30 minutes prior to having an ear temperature measurement taken.
* The subject exhibits symptoms of an acute or chronic inflammatory condition of the external ear canal. An example would be swimmer's ear. The subject may be included if the acute or chronic inflammatory condition is isolated to one ear, then the other ear may be used for data collection.
* The subject has an ear obstruction or excess cerumen build-up.
* The subject is in acute distress, i.e., severe pain, severe emotional distress or agitation that would inhibit them from participating in a tympanic ear temperature study.
* The subject has any known contraindication to oral, ear, or axillary temperature measurements.
* The subject has used ear drops in the last 8 hours. The subject may be included if the other ear was not medicated with ear drops in the last 8 hours.
* The subject (age 5+) has consumed food or drink, or smoked, within the last 20 minutes. The subject may be included if they wait 20 minutes prior to taking oral temperature.
* The subject has taken an antipyretic (ex: Tylenol, Motrin, Aspirin) in the last 120 minutes.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects recruited to participate in this study may range in age from normal weight (≥2.5kg), full-term (37 weeks gestation) newborns to geriatric adults. The subject may be anyone who is willing to have their temperature taken who also meets the eligibility criteria. Study subjects may have normal, febrile, or cold temperatures.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Bias | Immediately after the diagnostic test
  The mean difference between output temperatures of the clinical thermometer under test

SECONDARY OUTCOMES:
Repeatability | Immediately after the diagnostic test
  Pooled standard deviation (over a selected group of subjects) of changes in multiple output temperatures taken from the same subject at the same measuring site with the same clinical thermometer by the same operator within a relatively short time
Limits of Agreement | Immediately after the diagnostic test
  The magnitude of a potential disagreement between outputs of two clinical thermometers equal to double the standard deviation of output temperature differences when used on the same human subject.

CONTACTS AND LOCATIONS:
Locations (1):
- Baxter, Skaneateles, New York, United States

IPD SHARING:
Plan to Share IPD: No